CLINICAL TRIAL: NCT05546489
Title: A Proof-of-concept Study of Lymfit: A Personalized, Virtual Exercise Intervention to Improve Health Outcomes in Lymphoma Survivors in the Pandemic
Brief Title: Proof-of-concept Lymfif
Acronym: QI_LF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Christine Maheu, Associate Professor, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: QI_LF
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Quality of Life
Keywords: Quality of Life; cancer survivors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lymfit intervention (Experimental): Participants will receive a Fitbit wearable tracker, expert guidance, and a personalized exercise prescription to optimize physical activities among lymphoma survivors. The intervention is 12 weeks long, participants are meeting with a kinesiologist every 2 weeks.
  Interventions: Behavioral: Lymfit intervention

INTERVENTIONS:
Behavioral: Lymfit intervention — Wearable activity trackers (Fitbit) were given to participants as a motivational tool and for data collection purposes. Participants received a personalized exercise prescription designed by a kinesiologist. Physiologic metrics were collected by the Fitbit monitors and were stored in the Lymfit database. Self-reported questionnaires measuring health outcomes were collected at baseline and post-intervention.

SUMMARY:
This proof-of-concept study was to explore the implementation feasibility to deliver the Lymfit intervention to participants remotely during the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* 1. previously diagnosed with lymphoma
* 2. have completed chemotherapy
* 3. had access to a smart phone or an electronic device (e.g., tablet) that allowed them to attend virtual meetings and install the Fitbit application

Exclusion Criteria:

-1. have any contra-indications to performing physical activities as determined by the hematologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life : changes from baseline to post-intervention | 12 weeks
  Patient-Reported Outcomes Measurement Information System 29 items The scale has 29 items which measure perceived health status along 7 domains (physical function, anxiety, depressive symptoms, fatigue, sleep disturbance, ability to participate in social roles and activities, and pain interference), with items answered on five-point Likert scales. Raw scores generated for each domain will be transformed into a T score. The T score range from -0.022 to 1.0, with higher scores indicating greater endorsement of the construct being assessed.

SECONDARY OUTCOMES:
Fear of Cancer Recurrence : changes from baseline to post-intervention | 12 weeks
  Fear of Cancer Recurrence Inventory 42 items
Fear related to the pandemic : changes from baseline to post-intervention | 12 weeks
  the Fear of 2019 coronavirus disease (COVID) scale 7 items The items are rated on a five-point Likert scale ranging from "strongly disagree" (1) to "strongly agree" (5) with total scores ranging from 7 to 35. Higher total scores represent higher levels of fear.

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No